CLINICAL TRIAL: NCT06563505
Title: A Phase 2 Trial of Mosunetuzumab and Zanubrutinib for Patients With Relapsed/Refractory Marginal Zone Lymphoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-0243; NCI-2024-06965 (Other: NCI-CTRP Clinical Trial Registry)
Record Dates: First submitted 2024-08-19; First posted 2024-08-20 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Lymphoma
MeSH Terms: conditions — Lymphoma | interventions — zanubrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment w/Mosunetuzumab + Zanubrutinib (Experimental)
  Interventions: Drug: Mosunetuzumab; Drug: Zanubrutinib

INTERVENTIONS:
Drug: Mosunetuzumab — Given by IV
  Other Names: RO7030816
Drug: Zanubrutinib — Given by IV

SUMMARY:
To assess the efficacy and safety of mosunetuzumab combined with zanubrutinib in patients with relapsed or refractory MZL.

DETAILED DESCRIPTION:
Primary Objectives:

To determine the safety and efficacy of mosunetuzumab in combination with zanubrutinib as determined by best complete response (CR) rate of combination treatment for patients with relapsed or refractory marginal zone lymphoma (MZL).

Secondary Objectives:

To determine best overall response rate (ORR), duration of response (DOR), time to next treatment, progression-free survival (PFS), overall survival (OS), and evaluation of tolerability of mosunetuzumab and zanubrutinib as treatment for patients with relapsed/refractory MZL.

Exploratory Objective:

To determine the impact of total metabolic tumor volume to ORR, CR rate and survival outcomes

To determine the biomarkers that correlates with response and mechanisms of resistance to mosunetuzumab and zanubrutinib in relapsed/refractory MZL.

To determine the surrogate endpoint for future trials in MZL.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet the following criteria for study entry:

1. Histologically diagnosed marginal zone lymphoma (any subtypes)

   o Low grade or indolent B-cell lymphoma unclassifiable is also eligible
2. Have received at least 1 prior treatment including CD20 monoclonal antibody
3. Patients have relapsed or refractory disease to their most recent regimen
4. Stage II, III or IV disease
5. Age ≥18 years. Because no dosing or adverse event data are currently available on the use of mosunetuzumab and zanubrutinib combination in patients <18 years of age, children are excluded from this study.
6. Performance status ≤2 on the ECOG scale (≤3 if due to lymphoma)
7. Requiring systemic therapy assessed by investigator based on tumor size, symptoms and/or GELF criteria

   * A nodal or extranodal (except spleen) mass > 7 cm in its greater diameter
   * At least 3 nodal or extranodal sites ≥ 3 cm in diameter
   * Presence of at least one B symptom
   * Fever (>38 C), night sweats, weight loss > 10% in the past 6 months
   * Symptomatic splenomegaly (or size >13cm)
   * Impending organ compression or involvement (ureteral, orbital, gastrointestinal)
   * Any of the following cytopenias due to bone marrow involvement of lymphoma

     * Hemoglobin ≤ 10 g/dL
     * Platelets ≤ 100 x 109/L
     * Absolute neutrophil count (ANC) < 1.5x109/L
   * Pleural effusion or ascites
   * LDH > ULN or β2 microglobulin > ULN
8. Bi-dimensionally measurable disease, with at least one nodal lesion ≥ 1.5 cm or one extra-nodal lesion > 1 cm in longest diameter by CT, PET/CT, and/or MRI

   * Subjects with splenic MZL who do not meet the radiographically measurable disease criteria are eligible for participation if spleen is enlarged over 16 cm and MZL is histologically confirmed by bone marrow biopsy or peripheral blood flow cytometry
   * Subjects with EMZL such as skin of conjunctival EMZL who do not meet the radiographically measurable disease criteria are eligible for participation if at least one of the skin lesions is histologically confirmed as MZL and measures ≥1.5 cm in diameter
9. Patients must have adequate organ and marrow function as defined below:

   * Total bilirubin ≤ 1.5 institutional ULN, unless consistent with Gilbert's (ratio between total and direct bilirubin > 5)
   * AST (SGOT) and ALT (SGPT) ≤ 3 x institutional ULN
   * Alkaline phosphatase < 2.5 ULN
   * Creatinine clearance ≥ 40 ml/min calculated by modified Cockcroft-Gault formula
   * Blood counts below if without lymphoma cause for cytopenia
   * Hemoglobin ≥ 8 g/dL
   * Platelets ≥ 75 x 109/L
   * Absolute neutrophil count (ANC) ≥ 1.0x109/L
   * Blood counts below if cytopenia are due to lymphoma (such as bone marrow involvement or splenomegaly)

     * Hemoglobin ≥ 6 g/dL (no transfusion within 7 days prior to treatment)
     * Platelets ≥ 50 x 109/L
     * Absolute neutrophil count (ANC) ≥ 0.5x109/L

Exclusion Criteria:

Subjects will be ineligible for this study if they meet any of following criteria:

1. Known active central nervous system lymphoma or leptomeningeal disease.
2. Treatment with any chemotherapeutic agent, or treatment with any other anti-lymphoma agent (investigational or otherwise) within 4 weeks or five half-lives of the drug, whichever is shorter, prior to first investigational agent administration.
3. Any prior history of other malignancy besides B-NHL, unless the patient has been free of disease for ≥ 3 years and felt to be at low risk for recurrence by the treating physician, except:

   * Adequately treated localized skin cancer without evidence of disease.
   * Adequately treated cervical carcinoma in situ without evidence of disease.
4. Any life-threatening illness, medical condition, or organ system dysfunction which, in the investigator's opinion, could compromise the subject's safety, interfere with the absorption or metabolism of lenalidomide capsules, or put the study outcomes at undue risk.
5. Uncontrolled human immunodeficiency virus (HIV), or active Hepatitis C Virus, or active Hepatitis B Virus infection, or any uncontrolled active significant infection, including suspected or confirmed JC virus infection and SARS-CoV2.
6. Patients with inactive hepatitis B infection must adhere to hepatitis B reactivation prophylaxis unless contraindicated. Hepatitis B or C serologic status: subjects who are hepatitis B core antibody (anti-HBc) positive and who are surface antigen negative will need to have a negative polymerase chain reaction (PCR). Those who are hepatitis B surface antigen (HBsAg) positive or hepatitis B PCR positive will be excluded. Subjects who are hepatitis C antibody positive will need to have a negative PCR result. Those who are hepatitis C PCR positive will be excluded. Subjects with a history of Hepatitis C who received antiviral treatment are eligible as long as PCR is negative.
7. History of immunodeficiency (with the exception of hypogammaglobulinemia) or concurrent systemic immunosuppressant therapy (e.g., cyclosporine, tacrolimus, etc., or chronic administration glucocorticoid equivalent of >10mg/day of prednisone) within 28 days of the first dose of study drug with exception of steroid used for IV contrast allergy. In addition, use of inhaled, topical, intranasal corticosteroids or local steroid injection (eg, intra- articular injection) is permitted.
8. Use of strong/moderate inhibitors within 7 days or 5 half-lives prior to the first dose of zanubrutinib; usage of strong/moderate CYP3A inducers within 14 days prior to the first dose of zanubrutinib.
9. Requiring ongoing therapy with strong or moderate CYP3A inducers.
10. Clinically significant cardiovascular disease such as uncontrolled or symptomatic arrhythmias, congestive heart failure, or myocardial infarction within 6 months of Screening, or any Class 3 (moderate) or Class 4 (severe) cardiac disease as defined by the New York Heart Association Functional Classification. Subjects with controlled, asymptomatic atrial fibrillation during screening can enroll on study.
11. Significant screening electrocardiogram (ECG) abnormalities including 2nd degree atrioventricular (AV) block, type II AV block, or 3rd degree block.
12. Active bleeding or known bleeding diathesis (e.g., von Willebrand's disease) or hemophilia.
13. History of stroke or intracranial hemorrhage within 6 months prior to study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-12-11 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety and Adverse Events (AEs) | Through study completion; an average of 1 year.
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Dai Chihara, MD,PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org